CLINICAL TRIAL: NCT06007807
Title: Registry of Patients With Severe Trauma Admitted to the ICU in Tarragona
Brief Title: Severe Trauma Registry in Tarragona
Acronym: IcuTrauma
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Principal Investigator, Gerard Moreno, PhD, Staff of Intensive Care Unit, Hospital Universitari Joan XXIII de Tarragona.
Other Study IDs: ICUTRAUMA
Record Dates: First submitted 2023-08-04; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Major Trauma; Traumatic Brain Injury
Keywords: Severe trauma; Traumatic Brain Injury; ICU; Mortality; Trauma-induced coagulopathy; Hemorrhage
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe trauma is one of the leading causes of morbidity, mortality, and disability worldwide. Currently, it is the primary cause of death among individuals under 45 years of age. This disease, considered a "silent pandemic," exhibits heterogeneous physiopathology and unequal geographic distribution in terms of the type of injuries. The prognosis of subjects who have suffered severe trauma is uncertain, especially in patients with traumatic brain injury.

The epidemiology of severe trauma has undergone changes in recent years due to the global aging of society, resulting in different populations with older ages and more associated comorbidities. These factors are frequently linked to the use of chronic treatments such as antiplatelet agents or anticoagulants, which could worsen traumatic hemorrhage-the leading preventable cause of death following severe trauma. Despite efforts for primary prevention, such as road safety campaigns and occupational risk prevention, the annual incidence of severe trauma cases worldwide remains high. Enhancing the management of trauma patients would significantly influence the final clinical outcomes.

Given the aforementioned, it is of vital importance to understand the local epidemiology of severe trauma for the development of clinical research. This constitutes an effective tool to investigate changes in clinical practices, improve prevention strategies, and determine the global burden of the disease.

The hypothesis of the IcuTrauma Project is to create a territorial Registry of adults with severe trauma admitted to the ICU to understand the local epidemiology in Tarragona (Spain). This initiative would facilitate new lines of clinical research aimed at improving outcomes and the quality of care for trauma patients.

DETAILED DESCRIPTION:
* Study design: observational, retrospective, one centre (Hospital Universitari Joan XXIII) in Tarragona, Catalonia, Spain.
* Study period: Seven-years period: Since 01 January 2015 - 31 December 2022 (The registry will be open and active recruiting after this time point).
* Sample size calculation: Not applicable. The sample size will be equal to the total number of patients consecutively admitted to the Intensive Care Unit (ICU) due to severe trauma during the study period.
* Data extraction:

Data will be extracted by twofold:

1. Hand-driven: extracted data from the medical reports by reviewing the clinical history system performed by the study investigators, who are part of the staff of the ICU involved in the care of trauma patients. This information was collected into a large-scale database and, once introduced, the data was checked and verified by two investigators (and principal investigator).

   These manually extracted data included pre-hospital variables (such as the time of the injury, the mechanism of injury, first vital signs, pre-hospital procedures), in-hospital information (demographic's, primary survey of trauma in emergency department-ED, use of Extended Focused Assesment with Sonography in Trauma, complete laboratory results in ED), description of detailed anatomic injuries (Traumatic Brain Injury-TBI, thoracic trauma, abdominal trauma, Pelvic trauma, orthopedic injuries), severity scores (Acute Physiology And Chronic Health Evaluation-APACHE II, Sequential Organ Failure Assessment-SOFA score, Injury Severity Score-ISS, Abbreviated Injury Score-AIS, etc), resources during ICU admission (surgeries, transfusions, organ support, etc), complications (organ failures and nosocomial infections such as ventilator-associated pneumonia, catheter-related infection, etc), and clinical outcomes (ICU mortality, cause of death, in-hospital mortality, one-year survival, mechanical ventilation days, ICU and hospital length of stay, disability at ICU discharge and destination at discharge.
2. Automatic data: automated data collected with the Electronic Health System (Centricity Critical Care) provide solid and valid extraction of information. Automatic variables were checked and validated by the expert and specialized members of the ICU in data quality assessment and the management of data to ensure that recorded information was reliable. The accuracy, completeness and representativeness of automatic data was double checked when entered into the large-scale database for data quality by the principal investigator and a biotechnologist, who were responsible for the quality assurance plan that addressed data validation, monitoring and auditing (identifying inconsistencies, outliers or incorrect ranges for variables entered into the registry). The automated variables collected (not recorded manually) included demographic data, comorbidities and previous risk factors, dates (hospital and ICU admission, hospital and ICU discharge), laboratory tests during the first week of ICU admission, resources consumption during ICU stay, complications during ICU admission and outcomes.

   * Statistical plan: descriptive and analytical statistics using binary logistic regression (for association), survival analysis with Kaplan Meier analysis and Cox regression (for clinical outcomes), nonlinear association test such as CHAID decision analysis and restricted cubic splines, and matching learning analysis (for cluster or subgroups identification). These analyzes will be carried out using SPSS v24 and R software. Missing data values of automated variables will be handled using multiple imputation. Hand-driven data had negligible missing values.
   * Variable definitions (all definitions met the ATLS-Advanced Trauma Life Support criteria):

     * Previous anticoagulants or antiplatelet agents: chronic use of aspirin, clopidogrel, other antiplatelet agents, acenocumarol, warfarin, new anticoagulants.
     * Pre-hospital airway protection: includes supraglottic device, orotracheal intubation or surgical airway protection.
     * Penetrating trauma: knifes, firearm, impalement or others.
     * Flail chest: more than 3 ribs with fracture in two points.
     * Lung contusion: pulmonary infiltrate or condensation on initial X-rays after trauma.
     * Hemothorax type: simple (any pleural fluid detected after trauma), massive (>1.5 Liters acute or > 200cc/h in 2-4 hours).
     * Type of pneumothorax: simple (presence of aire in pleural space), hypertensive (with hypotension and/or respiratory failure).
     * Myocardial dysfunction (ventricular dysfunction detected in echocardiography or worsening of previous cardiac dysfunction).
     * Abdominal injuries grade (hepatic, spleen and renal trauma): anatomical scale injury using the AAST-The American Association for the Surgery of Trauma.
     * Pelvic fracture classification: Young-Burgees pelvic ring injury classification.
     * Neurogenic shock: bradycardia with hypoperfusion.
     * Urgent surgery: first 24 hours after trauma.
     * Hemorragia shock: hypoperfusion (with or without hypotension) defined by tachicardia, coldness, peripheral vasoconstriction, need for vasopressors, altered mental status, oliguria, hyperlactatemia or base excess deficit < - 6 due to the loss of blood after injury.
     * Damage control surgery: Non-definitive surgery consisting in packing for hemorrhage control, open abdomen, intestinal contamination control.
     * Massive hemorrhage: >10 CH in the first 24 hours, life-threatening hemorrhage, or > four blood products in the first 2 hours after admission.
     * Intracranial hypertension (ICH): episode of Intracranial pressures > 20-22 mmHg maintained for more than five minutes.
     * First level of ICH measures: general measures, sedation, neuromuscular blockade, ventricular drainage, osmotherapy.
     * Second level of ICH measures: decompressive craniectomy or brabiturics administration.
     * Osmotherapy: administration of hypertonic saline or mannitol during admission.
     * Intracranial rebleeding: increase in hematoma volume from initial tomography (CT scan).
     * Organ donor: organ donation.
     * ARDS (Acute respiratory distress syndrome): according the Berlin criteria.
     * Protective mechanical ventilation: applying tidal volumes 6-8 ml/Kg ideal body weight.
     * Free liquid CT: neither solid nor hollow viscera injury.
     * Non-operative management (NOM) for abdominal trauma: solid organ injury detected in CT scan managed through conservative management (no need for surgery at least 6-8 hours).
     * MNO failure: urgent laparotomy after deciding NOM.
     * White laparotomy: absence of lesions observed in the laparotomy.
     * Abdominal compartment syndrome: results from the progression of steady-state pressure within the abdominal cavity to a repeated pathological elevation of pressure above 20mmHg with associated organ dysfunction.
     * Early MODS (Multiorgan dysfunction syndrome): dysfunction of two or more organs in the first 72 hours after trauma.
     * Renal failure: according to AKIN guidelines.
     * Trauma-induced Coagulopathy (TIC): prolongation of the prothrombin and activated partial thromboplastin times over 1.5 times the control values, or fibrinogen < 150 mg/dL or thrombocytopenia < 100.000/ml in the first 72 hours after trauma.
     * Septic shock: identification of sepsis plus organ failure or tissue hypoperfusion.
     * Thrombosis: any type (deep vein thrombosis, arterial, pulmonary embolism).
     * Tracheostomy: percutaneous or surgical.
     * Nosocomial infection: any infection diagnosed after 48 hours of ICU admission.
     * VAP (Ventilator-associated pneumonia): clinical and microbiologically confirmed pneumonia in patients ventilated for at least 48 hours.
     * VAT (Ventilator-associated tracheobronchitis): upper respiratory tract infection (without pneumonia) in patients ventilated for at least 48h.
     * CRI (Catheter-related infection): bacteremia with positive catheter culture for the same microorganism and no other source of infection, with a minimum of 15 colony formation units in the catheter culture.
   * Intra-abdominal infection: peritonitis, abscess, positive surgical fluid.
   * Infection of open fractures: positive culture of the wound.
   * MDR (multidrug resistant) infection: includes any bacteria resistant to at least three antibiotic families.
   * Limitation of life support: withholding or withdrawal.
   * Causes of death: hemorrhagic shock, early MODS, late MODS, septic shock, refractory ICH (without response to applied measures), others.

ELIGIBILITY:
Inclusion Criteria:

* Adults who were consecutevely admitted to the ICU for severe trauma during the study period.

Exclusion Criteria:

* Children aged < 15 years old.
* Trauma admitted outside the ICU

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting a severe trauma in the province of Tarragona and transferred to the Joan XXIII Hospital (Tarragona City), either as primary or secondary transfer. The ICUTRAUMA project was conducted in one center (Joan XXIII University Hospital), which is the reference center in the province. It is a Level II Trauma Center. It has 24-hours neurosurgery and ICU availability, being the reference centre in the province for patients with TBI. The Joan XXIII Hospital receives patients with severe trauma from other six centers. The entire province covers a total surface area of 6,302 km2 with almost 1M inhabitants. According to our general data, more than 400 patients are admitted to the hospital emergency department each year, of which more than 100 patients require admission to the ICU.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
ICU mortality | Time (in days) between ICU admission date and ICU discharge date
  proportion of deaths

SECONDARY OUTCOMES:
Length of stay (LOS) | Time (in days) between hospital admission date and hospital discharge date
  Hospital length of stay
Mechanical ventilation duration | During the invasive mechanical ventilation treatment
  Total duration and Ventilator-free days
In-hospital mortality | at 28 day
  Proportion of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Moreno, PhD, Principal Investigator — Hospital Universitari Joan XXIII
Locations (1):
- Hospital Universitari Joan XXIII, Tarragona, Catalonia/Tarragona, Spain